CLINICAL TRIAL: NCT02993744
Title: Assessment of Maternal Inflammatory Parameters Within Routine Treatment With Betamethasone Under Threat of Preterm Delivery
Brief Title: Maternal Inflammatory Parameters Within Routine Treatment With Betamethasone
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kastanek Maria, Student, Medical University of Vienna
Other Study IDs: 2130/2015
Record Dates: First submitted 2016-12-07; First posted 2016-12-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Preterm Birth
Keywords: preterm birth; corticosteroids; inflammatory parameters; betamethasone; leukocytes
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — - blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Group: 75 woman between the age of 18 to 50 years, week of gestation 23+0 - 34+6, threatening preterm delivery, application of Betamethasone
- Control Group: 65 woman between the age of 18 to 50 years, week of gestation 23+0 - 34+6, no threatening preterm delivery

SUMMARY:
It is the aim of this study to detect the effect of Betamethasone on the maternal inflammatory parameters C-reactive protein (CRP) and leukocytes of a pregnant woman under threat of preterm delivery, for example because of a cervical infection.

DETAILED DESCRIPTION:
BACKGROUND

Cortisone influences the maternal number of leukocytes and CRP of a pregnant woman. Because of that, it is difficult to know if the medical treatment of an infection was successful and accordingly if the diagnosis was justified.

METHODS

In this study, the blood results of 75 pregnant women under threat of preterm delivery (week of gestation 23+0 to 34+6), treated with Betamethasone will be analysed. 65 pregnant women without complications serve as control group.

ELIGIBILITY:
Inclusion Criteria:

* week of gestation 23+0 until 34+6

Exclusion Criteria:

* infectious diseases f.e. hepatitis B or C, HIV
* diseases of the thyroid gland

  75 Patients facing preterm labour 65 Patients acting as a control group, without preterm labor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant woman admitted to the department of feto-maternal health and obstetrics
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
CRP | 48h
  The CRP values in mg/dL before and 48h after the first Betamethasone application

SECONDARY OUTCOMES:
Leucocytes | 48h
  The Leucocyte values in G/L before and 48h after the first Betamethasone application

OTHER OUTCOMES:
Body Mass Index (BMI) | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  Body Mass Index (BMI) in kg/m^2 is calculated to test for influence on inflammatory parameters in both groups (case and control)
Weight | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  Weight in kilogram (kg) is taken from the medical record to calculate the BMI in both groups (case and control)
Height | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  Size in meters (m) is taken from the medical record to calculate the BMI in both groups (case and control)
CRP Control Group | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  CRP values in mg/dL of patients belonging to the control group
Leucocytes Control Group | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  Leucocyte values in G/L of patients belonging to the control group
Patients with Allergies | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  information about the patients allergie status (allergies yes or no) is taken from the medical record to test for influence on inflammatory parameters in both groups (case and control)
Patients with Diabetes | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  information about the patients diabetes status (diabetes yes or no) is taken from the medical record to test for influence on inflammatory parameters in both groups (case and control)
Smoking Habits | single point in the time frame between week of gestation 23+0 - 34+6, no fixed day
  information about the patients smoking status (smoking yes or no) is taken from the medical record to test for influence on inflammatory parameters in both groups (case and control)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kastanek, Principal Investigator — Medical University Vienna; Florian Frommlet, DI. Dr., Study Chair — Medical University Vienna
Locations (1):
- General Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No